CLINICAL TRIAL: NCT00705978
Title: A One Week Double-Blind, Randomized, Placebo-Controlled, Parallel Group, Multi-Center Study With Creon 40,000 MMS in Subjects With Pancreatic Exocrine Insufficiency Due to Chronic Pancreatitis, Followed by an Open-Label Long-Term Extension
Brief Title: Creon 40,000 for Treatment of PEI (Pancreatic Exocrine Insufficiency) Due to Chronic Pancreatitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott Products (Industry)
Collaborators: Datamap (Industry)
Responsible Party: Gregor Eibes, Clinical Trial Manager, Abbott Products
Organization: Abbott (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: S245.4.009
Record Dates: First submitted 2008-06-26; First posted 2008-06-27 (Estimated); Last update posted 2011-08-18 (Estimated); Status verified 2011-08

CONDITIONS: Pancreatic Insufficiency
Keywords: Pancreatic Exocrine Insufficiency Due to Chronic Pancreatitis
MeSH Terms: conditions — Exocrine Pancreatic Insufficiency | interventions — Pancreatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Pancreatin
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pancreatin — Pancreatin with 40000 lipase units per capsule, 2 capsules per main meal (3 main meals) plus 1 capsule per snack (2-3 snacks)
  Arms: 1
Drug: Placebo — placebo
  Arms: 2

SUMMARY:
This study will provide efficacy data for Creon 40,000 in CP subjects as well as long-term safety data. During the long-term treatment with Creon 40,000 nutritional parameters will be assessed and correlated with CFA.

ELIGIBILITY:
Inclusion Criteria

* Pancreatic exocrine insufficiency has to be proven (in medical history) by a pancreatic function test
* Chronic pancreatitis has to be proven (in medical history) by CT, ERCP, plain film with pancreatic calcifications, ultrasonography (calcifications,duct dilatation) and /or histology
* Females must be non-lactating and either be of non-childbearing potential or if of childbearing potential, agree to practice effective barrier contraceptive methods, use an intrauterine device (IUD) or use birth control pills or equivalent injectable contraceptive. The subject must have been practicing the selected method of birth control for at least 3 months prior to Visit 1 (Day -14).
* Subjects with a pathological stool fat during run in period (> 10g/24 h)

Exclusion Criteria

* Ileus or acute abdomen
* Any type of malignancy involving the digestive tract in the last 5 years
* Presence of pseudo pancreatic cysts >= 4 cm
* Current excessive intake of alcohol or drug abuse
* Hypersensitivity vs porcine proteins / pancreatin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2008-06; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Change in CFA from baseline to the end of double blind treatment | 7 days after baseline

SECONDARY OUTCOMES:
CNA, stool fat, stool weight, nutritional, clinical symptomatology, SF-36, BMI | 7 days after baseline, and end of open-label period (1 year of open label treatment)

CONTACTS AND LOCATIONS:
Overall Officials: Guenter Krause, MD, Study Director — Abbott Products
Locations (11):
- India (11):
  - Site Reference ID/Investigator# 45389, Bangalore
  - Site Reference ID/Investigator# 45396, Bhopal
  - Site Reference ID/Investigator# 45390, Chennai
  - Site Reference ID/Investigator# 45391, Hyderabad
  - Site Reference ID/Investigator# 45388, Jaipur
  - Site Reference ID/Investigator# 54382, Kochi
  - Site Reference ID/Investigator# 45387, Kolkata
  - Site Reference ID/Investigator# 45383, Mumbai
  - Site Reference ID/Investigator# 45382, Pune
  - Site Reference ID/Investigator# 45395, Pune
  - Site Reference ID/Investigator# 45393, Trivandrum